CLINICAL TRIAL: NCT01789177
Title: Use of Disposable Spirometer for Recovery of Pulmonary Function by Peak Expiratory Flow Measurement Following Exploratory Laparotomy
Brief Title: Use of Disposable Spirometer for Recovery of Pulmonary Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-0055
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2014-03

CONDITIONS: Postoperative Complications
Keywords: Spirometry; Postoperative Care
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified incentive spirometry (Experimental): Patients will be given a disposable incentive spirometer postoperatively and instructed to use the spirometer every hour while awake.
  Interventions: Device: Incentive Spirometry; Other: Postoperative chest physiotherapy
- Postoperative chest physiotherapy (Active Comparator): Patients will be given standard postoperative chest physiotherapy, according to hospital protocol, but will not receive incentive spirometers.
  Interventions: Other: Postoperative chest physiotherapy

INTERVENTIONS:
Device: Incentive Spirometry — Patients will be provided with plastic, disposable incentive spirometers postoperatively
  Arms: Modified incentive spirometry
Other: Postoperative chest physiotherapy — Patients will be given routine postoperative chest physiotherapy instruction by nursing staff

SUMMARY:
We hypothesize that the addition of modified incentive spirometry to standard postoperative chest physiotherapy will be associated with faster return to baseline/predicted pulmonary function and fewer postoperative pulmonary complications in patients following laparotomy.

DETAILED DESCRIPTION:
The primary objective of this study is to determine how quickly patients' peak expiratory flow measurement returns to baseline or predicted values following laparotomy with or without the assistance of modified incentive spirometry. The secondary objective is to assess the effectiveness of modified incentive spirometry in preventing postoperative pulmonary complications in patients following laparotomy. Specifically, this study will track length of stay, mortality, and evidence of pulmonary infection in both treatment and non-treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who undergo laparotomy at Kamuzu Central Hospital, Malawi

Exclusion Criteria:

* Patients with known pre-existing pulmonary disease
* Pregnant women
* Patients who cannot perform maximal expiration for measurement of peak expiratory flow meter because of inability to understand or follow directions and demonstrations
* Patients with terminal cancer or illness with life-expectancy less than 1 month
* Patients with burn injuries
* Patients with illness requiring intubation and mechanical ventilation or postoperative ICU admission
* Patients who require additional operations during the course of their hospital stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Return to baseline or predicted pulmonary function | postoperative course up to discharge
  Return to baseline/predicted pulmonary function based on peak expiratory flow measurement. Postoperative measurement will be compared to preoperative measurement (for elective cases) or age-predicted measurement (for emergency cases)

SECONDARY OUTCOMES:
Incidence of postoperative pulmonary complications | postoperative course until discharge
  We will measure length of hospital course, mortality, and incidence of pneumonia, pleural effusion, or other postoperative pulmonary complication based on clinical diagnosis and available radiological studies

CONTACTS AND LOCATIONS:
Overall Officials: Anthony G Charles, MD, Principal Investigator — UNC Department of Surgery
Locations (1):
- Kamuzu Central Hospital, Lilongwe, Malawi

REFERENCES:
- [Background] Brooks-Brunn JA. Postoperative atelectasis and pneumonia. Heart Lung. 1995 Mar-Apr;24(2):94-115. PMID 7759282
- [Background] Canet J, Mazo V. Postoperative pulmonary complications. Minerva Anestesiol. 2010 Feb;76(2):138-43. Epub 2009 Nov 24. PMID 20150855
- [Background] Ferreyra G, Long Y, Ranieri VM. Respiratory complications after major surgery. Curr Opin Crit Care. 2009 Aug;15(4):342-8. doi: 10.1097/MCC.0b013e32832e0669. PMID 19542885
- [Background] Ferreyra GP, Baussano I, Squadrone V, Richiardi L, Marchiaro G, Del Sorbo L, Mascia L, Merletti F, Ranieri VM. Continuous positive airway pressure for treatment of respiratory complications after abdominal surgery: a systematic review and meta-analysis. Ann Surg. 2008 Apr;247(4):617-26. doi: 10.1097/SLA.0b013e3181675829. PMID 18362624
- [Background] Lawrence VA, Cornell JE, Smetana GW; American College of Physicians. Strategies to reduce postoperative pulmonary complications after noncardiothoracic surgery: systematic review for the American College of Physicians. Ann Intern Med. 2006 Apr 18;144(8):596-608. doi: 10.7326/0003-4819-144-8-200604180-00011. PMID 16618957
- [Background] Restrepo RD, Wettstein R, Wittnebel L, Tracy M. Incentive spirometry: 2011. Respir Care. 2011 Oct;56(10):1600-4. doi: 10.4187/respcare.01471. PMID 22008401
- [Background] Westwood K, Griffin M, Roberts K, Williams M, Yoong K, Digger T. Incentive spirometry decreases respiratory complications following major abdominal surgery. Surgeon. 2007 Dec;5(6):339-42. doi: 10.1016/s1479-666x(07)80086-2. PMID 18080608
- [Derived] Tyson AF, Kendig CE, Mabedi C, Cairns BA, Charles AG. The effect of incentive spirometry on postoperative pulmonary function following laparotomy: a randomized clinical trial. JAMA Surg. 2015 Mar 1;150(3):229-36. doi: 10.1001/jamasurg.2014.1846. PMID 25607594